CLINICAL TRIAL: NCT05889988
Title: A Study of the Natural History of Ado-trastuzumab Emtansine (T-DM1)-Induced Peripheral Neuropathy in HER2-positive Breast Cancer Patients
Brief Title: A Study of Ado-trastuzumab Emtansine (T-DM1)-Induced Peripheral Neuropathy in HER2-positive Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC220904; 22-010634 (Other: Mayo Clinic Institutional Review Board); MNCCTN031 (Other: Minnesota Cancer Clinical Trials Network)
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasm
Keywords: Ado-trastuzumab emtansine (T-DM1); Peripheral Neuropathy; HER2-positive
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2 Metastatic Group: HER2 Metastatic Setting (defined by breast cancer that has spread outside of the breast and the immediately draining lymph node regions; stage IV)
- HER2 Adjuvant Group: HER2 Adjuvant Setting (defined by breast cancer that is not known to have spread outside of the breast and the immediately draining lymph node regions; stages I-III). The Adjuvant Setting includes patients receiving neoadjuvant therapy.

SUMMARY:
Researchers plan to study the natural history of ado-trastuzumab emtansine (T-DM1)-induced neuropathy both in patients without any history of neuropathy or previous neurotoxic agent use and in patients who have such a history.

ELIGIBILITY:
Inclusion Criteria:

* Planning to receive three or more doses T-DM1 for HER2-positive metastatic breast cancer (any line) or for earlier-stage breast cancer. The patient may have received one dose of T-DM1, prior to study entry if it has not been longer than 14 days since that dose and that the patient will be able to complete the required baseline questionnaire within 14 days of their first dose of T-DM1.
* Patients with previous use of neurotoxic antineoplastic agents (excluding previous use of T-DM1), pre-existing CIPN, or peripheral neuropathy secondary to other causes will be able to be enrolled in the study.
* The patient plans to continue clinical follow-up at the same institution, where the patient entered the study.
* Provide informed consent.
* Ability to complete questionnaire(s) in English by themselves or with assistance.

Exclusion Criteria:

* Previous use of T-DM1
* Concomitant use of other neurotoxic anticancer agents including cisplatin, carboplatin, oxaliplatin, docetaxel, paclitaxel, vincristine, eribulin, vinorelbine, thalidomide, lenalidomide, bortezomib, or epothilones. If the patient used any of these previously, then they must have been stopped for at least 7 days prior to study entry.
* Current use of commonly used drugs for the treatment of peripheral neuropathy, including duloxetine, gabapentinoids (pregabalin and gabapentin), venlafaxine, nortriptyline, or amitriptyline (including use of these medications for things other than neuropathy). If the patient used any of these previously, then they must have been stopped for at least 7 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients planning to receive three or more doses of Ado-trastuzumab emtansine (T-DM1) for HER2-positive metastatic breast cancer or for earlier-stage breast cancer. Patients must have previously used neurotoxic antineoplastic agents (excluding previous use of T-DM1), have pre-existing chemotherapy-induced peripheral neuropathy (CIPN), or have peripheral neuropathy secondary to other causes. Patients must also plan to continue clinical follow-up at the same institution where they enter the study.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in chronic neuropathy symptoms | Baseline, approximately 22 months
  Measured using the European Organisation of Research and Treatment of Cancer Quality of Life Questionnaire-Chemotherapy-induced peripheral neuropathy (CIPN) twenty-item scale (EORTC QLQCIPN20), a validated instrument designed to elicit cancer patients' experience of symptoms and functional limitations related to chemotherapy-induced peripheral neuropathy. The total score of CIPN20, each of the three subscale scores (sensory, motor, autonomic), and each individual item of the CIPN20 tool will be computed following standard scoring algorithm and converted into a 0-100 scale; higher scores indicate greater severity of neuropathy symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dan S. Childs, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (21):
- United States (21):
  - Riverwood Healthcare Center, Aitkin, Minnesota
  - Essentia Health Baxter Clinic, Baxter, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Ely Clinic, Ely, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Fairview Grand Itasca Clinic & Hospital, Grand Rapids, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Fairview Range Medical Center, Hibbing, Minnesota
  - Essentia Health - International Falls Clinic, International Falls, Minnesota
  - MMCORC CentraCare Monticello Cancer Center, Monticello, Minnesota
  - Essentia Health Moose Lake, Moose Lake, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Health Thief River Falls Clinic, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Health Worthington, Worthington, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials